CLINICAL TRIAL: NCT01395199
Title: Amlodipine in the Prevention and Treatment of Iron Overload in Patients With Thalassemia Major: a Randomized, Controlled Trial
Brief Title: Amlodipine in the Prevention and Treatment of Iron Overload in Patients With Thalassemia Major
Acronym: AmloThal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Juliano de Lara Fernandes, Physician Researcher, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AmloThal RCT
Record Dates: First submitted 2011-07-11; First posted 2011-07-15 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Thalassemia; Iron Overload
Keywords: Magnetic resonance imaging; Thalassemia; Iron overload
MeSH Terms: conditions — Thalassemia; Iron Overload | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Starch pill (Placebo Comparator): Placebo
  Interventions: Drug: Amlodipine
- Amlodipine (Experimental): Amlodipine 5mg QD
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — 5mg PO initially; may be reduced to 2.5mg PO if side effects
  Other Names: norvasc

SUMMARY:
This study aims to investigate the use of amlodipine, a drug that blocks the uptake of calcium into cells, in the prevention and treatment of iron overload in patients with thalassemia major. Since iron uses the same calcium channels to enter the heart, pancreas and other organs, blocking these channels might help to prevent the accumulation of iron in these tissues. The study will follow 60 patients with thalassemia major: 30 will receive amlodipine and 30 will serve as controls receiving placebo in a randomized double-blind fashion. Patients will be monitored through one year. Monitoring will occur through the measurement of blood ferritin as well as live and heart T2* by MRI initially, at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thalassemia major with at least 6 years of age undergoing iron chelation therapy.
2. No anticipated changes in chelation regimen for the next 12 months
3. Completed and signed Informed Consent

Exclusion Criteria:

1. Pregnancy
2. Advanced class III/IV heart failure or LVEF < 0.35% (by MRI)
3. Formal contra-indications to MRI (pacemakers, cerebral aneurysm metal clips, etc).
4. Advanced heart AV block

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Myocardial T2* values (msec) | 6 and 12 months
  T2* values represent the amount of iron in the myocardial and is quantified in msec and measured by cardiovascular magnetic resonance

SECONDARY OUTCOMES:
Liver T2* values (msec) | 6 and 12 months
  T2* values represent the amount of iron in the liver and is quantified in msec and measured by cardiovascular magnetic resonance
Serum ferritin levels | 6 and 12 months
left ventricle volumes and function | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juliano L Fernandes, MD, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Universidade Estadual de Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597
- [Derived] Fernandes JL, Loggetto SR, Verissimo MP, Fertrin KY, Baldanzi GR, Fioravante LA, Tan DM, Higa T, Mashima DA, Piga A, Coelho OR, Costa FF, Saad ST. A randomized trial of amlodipine in addition to standard chelation therapy in patients with thalassemia major. Blood. 2016 Sep 22;128(12):1555-61. doi: 10.1182/blood-2016-06-721183. Epub 2016 Jul 13. PMID 27412888
- See also: Brazilian Thalassemia Association — http://www.abrasta.org.br/